CLINICAL TRIAL: NCT00304421
Title: Comparison of the Nighttime Effects of Rabeprazole 20 mg to Pantoprazole 40 mg on Standard Meal Stimulated Gastric Acid Secretion and Intragastric pH in H. Pylori Negative Volunteer Subjects With GERD
Brief Title: Comparison of the Nighttime Effects of Two Different Drugs on Subjects With GERD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry); Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0028
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease; Proton Pump Inhibitors; Gastric pH; Gastric Acid Secretion
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole; Pantoprazole

INTERVENTIONS:
Drug: rabeprazole
Drug: pantoprazole

SUMMARY:
The purpose of the study is to compare the effect of two different drugs, rabeprazole (20 mg) and pantoprazole (40 mg), and their effects on the amount of acid produced by your stomach on evening and at night after standard protein meal.

DETAILED DESCRIPTION:
Gastric acid secretion can be divided into two phases: the daytime phase and the nocturnal phase. Nocturnal acid reflux is presumably more damaging because of loss of salivary neutralization. The present study is designed to measure effects of rabeprazole and pantoprazole on post-prandial and nocturnal gastric acid secretion and intragastric pH in H. pylori-negative volunteers with gastroesophageal reflux disease. These measurement will be used to compare the degree of inhibition of gastric acid secretion between the two drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, 18-65 years of age, inclusive, male or female, of any race, who are willing to undergo testing at the study center.
2. Female subjects must not be able to conceive by reason of surgery, radiation, 2 years past the onset of menopause, or an approved method of contraception (e.g., IUD, oral contraceptives for at least one cycle, implant, or double barrier method). Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test before medication is dispensed.
3. Subjects must have a negative result on the screening for H. pylori by serology, and no history of H. pylori eradication.
4. Subjects must have history of GERD with or without antacid use.
5. Subjects must be able to tolerate nasogastric tube placement.

Exclusion Criteria:

1. History of gastric surgery, fundoplication or vagotomy.
2. Pyloric stenosis Barrett's esophagus or esophageal stricture.
3. Treatment with a histamine H2-receptor antagonist, prostaglandin, or sucralfate within 14 days before enrollment into this study.
4. Treatment with rabeprazole, omeprazole, lansoprazole, pantoprazole, esomeprazole, prokinetic agent, or bismuth subsalicylate within 30 days before enrollment into this study.
5. Concurrent serious systemic disorders, including renal insufficiency and hepatic insufficiency.
6. Subjects with neoplasia or undergoing treatment for cancer (e.g., chemotherapy, radiation.
7. Any condition associated with poor subject compliance (e.g., alcohol abuse, drug abuse).
8. History of clinically significant abuse of alcohol defined as (1) patterns of alcohol intake consistent with disruption of normal function in society; (2) history of, or current existence of any indication of difficulty in abstaining from alcohol for the required duration of the present protocol; (3) use of any alcohol within one day of any study period.
9. Subjects who have received any investigational agent within the previous 30 days.
10. Inability of subject to return for scheduled visits.
11. Subjects who, in the opinion of the investigator, are poor medical or psychiatric risks for therapy with an investigational drug.
12. History of any hypersensitivity reaction to rabeprazole, pantoprazole or any of their inactive ingredients.
13. Any significant evidence at screening of endocrine, cardiovascular, and/or pulmonary disorder.
14. Any predisposing condition that might interfere with the absorption, distribution, metabolism, or excretion of drug, or a history of abnormal bleeding tendencies or thrombophlebitis.
15. History of HIV, hepatitis B, or hepatitis C infection.
16. Subjects who are pregnant or likely to become pregnant during the course of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2004-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that during the hours 2000 through 0800 following a single dose administration of medication, the median change from baseline values in gastric acid secretion with 20 mg rabeprazole is significantly less than 40 mg pantoprazole

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pisegna, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States